CLINICAL TRIAL: NCT01457612
Title: Effect of 6 Weeks Strawberry Supplementation on Insulin Action and Associated Risk Factors in Insulin Resistant (IR) Subjects (STR2)
Brief Title: Effect of 6-week Strawberry Supplementation on Insulin Action (STR2)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Nutrition Research Center, Illinois Institute of Technology (Industry)
Collaborators: California Strawberry Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STR2 2011-076
Record Dates: First submitted 2011-10-19; First posted 2011-10-24 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Insulin Resistance; Nutritional Disease; Metabolic Disease
Keywords: Insulin Resistant; Dietary Supplements; Nutrition; Antioxidant; Inflammation
MeSH Terms: conditions — Insulin Resistance; Nutrition Disorders; Metabolic Diseases; Inflammation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo1 (Placebo Comparator): Placebo Beverage 1 without fiber
  Interventions: Dietary Supplement: Placebo1
- Strawberry (Active Comparator): Strawberry Beverage 20g/BID
  Interventions: Dietary Supplement: Strawberry
- Placebo2 (Placebo Comparator): Placebo Beverage 2 with Fiber
  Interventions: Dietary Supplement: Placebo2

INTERVENTIONS:
Dietary Supplement: Strawberry — 20g twice per day (BID) in beverage
  Arms: Strawberry
Dietary Supplement: Placebo1 — Placebo Beverage 1 without fiber
  Arms: Placebo1
Dietary Supplement: Placebo2 — Placebo Beverage 2 with Fiber
  Arms: Placebo2

SUMMARY:
The primary study objective is to investigate the potential chronic beneficial effect of polyphenolics derived from strawberry on impaired insulin signaling in insulin resistant individuals through their ability to modulate oxidative- and inflammatory-markers that lead to devastating disease, including, but not limited to, diabetes and cardiovascular disease.

DETAILED DESCRIPTION:
This study is a single-center, randomized and single blinded, placebo-controlled, 6-week, parallel design study with follow-up to evaluate strawberry-associated chronic improvements in insulin action resulting in reduced whole body insulin resistance and improved glucose tolerance. This study will take approximately 11~12 weeks.

Subjects will follow an extremely limited polyphenolic diet throughout the duration of their participation in the study.

The limited diet will begin 7 days before the first study visit and end before the last study visit. Following the polyphenol-free 7-day run in period, at Week 0, subjects will be scheduled to return to the Center for sequence randomization, an Oral Glucose Tolerance Test (OGTT) as well as a Flow Mediated Dilation (FMD) procedure to measure endothelial function. Subjects will incorporate either one of tow Placebo Beverages (PBO1, n=15; PBO2, n=15) or Strawberry Beverage (STR, n=15, an optimal strawberry test dose of 40 g/d) into their diet daily for a period of 6 weeks. Subjects will consume randomly assigned beverage twice per day with their breakfast and dinner meals.

All subjects will be asked to come to the Center once a week where they will receive a week's supply of beverages. Additionally, fasting clinical and laboratory variables, anthropometrics, and vital sign measurements will be assessed at each bi-weekly visit at Week 3 and Week 5.

Participants will undergo the same procedures at the end of Week 6: fasting blood sample collection for analysis of insulin, glucose, oxidative and inflammatory markers, an OGTT to assess glucose handling, as well as a FMD procedure to assess endothelial function in response to 6 weeks of either the Placebo or Strawberry treatment.

Subjects will be required to visit the Center 4 weeks after the end of their intervention period (Week 10), at which time they will undergo their last anthropometrics and vital sign measurements, a 4 hour OGTT, and the FMD procedure.

ELIGIBILITY:
Inclusion Criteria:

* Must meet ONE or MORE of the criteria (1)-(5) associated with insulin resistance along with all other criteria listed (6)-(9):

  1. Blood glucose concentration between140-199 mg/dL at 2hr from OGTT.
  2. Elevated fasting glucose (110 mg/dL≤ Fasting blood glucose <126 mg/dL)
  3. Elevated fasting insulin (>75th percentile cutoff of 13.13 μU/mL)
  4. Insulin resistance defined by the homeostasis model assessment method of insulin resistance (HOMA-IR) (glucose [in millimoles per liter] × insulin [in microunits per milliliter]/22.5) values of at least 2.5.
  5. Waist circumference ≥ 110 cm because many epidemiology studies have been shown that waist circumferences may be related to insulin resistance.
  6. Nonsmokers
  7. Not taking any medications that would interfere with outcomes of the study, i.e. lipid lowering medications, anti-inflammatory drugs, or dietary supplements
  8. 18 years of age and older
  9. No clinical evidence of cardiovascular, metabolic, respiratory, renal, gastrointestinal or hepatic disease

Exclusion Criteria:

* Pregnant and/or lactating.

  * Allergy or intolerance to strawberries and dairy products.
  * Current regular consumption of strawberries is > 2 servings per day.
  * Fasting blood glucose ≥ 126 mg/dL. Subjects identified with elevated fasting blood glucose levels will be advised to contact their primary care physician for appropriate follow-up care.
  * Taking over the counter antioxidant supplements or other supplements that may interfere with the study procedures or endpoints.
  * Subjects with unusual dietary habits (e.g. pica).
  * Actively losing weight or trying to lose weight (unstable body weight fluctuations of > 5 kg in a 60 day period).
  * Excessive exercisers or trained athletes.
  * Subjects with documented atherosclerotic disease, inflammatory disease, diabetes mellitus, or other systemic diseases.
  * Addicted to drugs and/or alcohol.
  * Medically documented psychiatric or neurological disturbances.
  * Smoker (past smoker may be allowed if cessation is > 2 years).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-10-01 (Actual); Primary Completion 2012-12-01 (Actual); Study Completion 2013-03-01 (Actual)

PRIMARY OUTCOMES:
The chronic beneficial effect of polyphenolics from strawberry on impaired insulin signaling in insulin-resistant men and women | 10 weeks
  Subjects will be randomized to receive either one of beverages, Pbo1, Pbo2 or Str Beverage and consume randomly assigned beverage twice per day with their breakfast and dinner meals for 6 weeks. On visits at Wk0, Wk6, and Wk10, blood will be collected at 0h, and 1h, 2h, 3h and 4h time points following the 75 g glucose load (oral glucose tolerance test) and Flow Mediated Dilation (FMD) procedure will be performed as well.

SECONDARY OUTCOMES:
The chronic beneficial effect of polyphenolics from strawberry on oxidative- and inflammatory-markers in insulin-resistant men and women | 10 Weeks
  Samples of venous blood will be collected for measurement of oxidative and inflammatory markers (hs-CRP levels, LDL oxidation, Interleukin (IL)-6 and other inflammatory molecules, Total antioxidant levels of the blood)

CONTACTS AND LOCATIONS:
Overall Officials: Indika Edirisinghe, Ph.D, Principal Investigator — Institute for Food Safety and Health; Britt Burton-Freeman, Ph.D, Principal Investigator — Institute for Food Safety and Health
Locations (1):
- Clinical Nutrition Research Center, Chicago, Illinois, United States

REFERENCES:
- [Result] Burton-Freeman B, Linares A, Hyson D, Kappagoda T. Strawberry modulates LDL oxidation and postprandial lipemia in response to high-fat meal in overweight hyperlipidemic men and women. J Am Coll Nutr. 2010 Feb;29(1):46-54. doi: 10.1080/07315724.2010.10719816. PMID 20595645
- [Result] Edirisinghe I, Burton-Freeman B, Varelis P, Kappagoda T. Strawberry extract caused endothelium-dependent relaxation through the activation of PI3 kinase/Akt. J Agric Food Chem. 2008 Oct 22;56(20):9383-90. doi: 10.1021/jf801864t. Epub 2008 Sep 25. PMID 18816058